CLINICAL TRIAL: NCT04542681
Title: A Phase I, Single-Blind, Placebo-Controlled Study Evaluating the Cardiovascular Properties of MANP in African Americans With Hypertension
Brief Title: MANP in African Americans With Hypertension
Acronym: MANP-2
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was withdrawn and replaced by a larger study
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Paul M. McKie, M.D., Consultant, Mayo Clinic
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 17-007947
Record Dates: First submitted 2018-12-18; First posted 2020-09-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: The study is designed in 2 cycles. The first cycle subjects will receive Placebo (n=10) or MANP 2.5 ug/kg (n=20). In the second cycle subjects will receive MANP 5 ug/kg/ (n=10).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo - 1st Cycle (Placebo Comparator): Subjects will receive a single SQ injection of placebo (0.9% normal saline) (n=10)
  Interventions: Drug: Placebo - 1st Cycle
- MANP - 1st Cycle (Active Comparator): Subjects will receive a single SQ injection of 2.5 μg/kg MANP (n=10)
  Interventions: Drug: MANP - 1st Cycle
- MANP - 2nd Cycle (Active Comparator): Subjects will receive a single SQ injection of 5 μg/Kg MANP (n=10)
  Interventions: Drug: MANP - 2nd Cycle

INTERVENTIONS:
Drug: Placebo - 1st Cycle — Subjects will receive a single SQ injection of placebo/normal saline
  Other Names: 0.9% Normal Saline
  Arms: Placebo - 1st Cycle
Drug: MANP - 1st Cycle — Subjects will receive a single SQ injection of MANP at a concentration of 2.5 μg/kg
  Other Names: Mutant ANP
  Arms: MANP - 1st Cycle
Drug: MANP - 2nd Cycle — Subjects will receive a single SQ injection of MANP 5 μg/kg concentration.
  Other Names: Mutant ANP
  Arms: MANP - 2nd Cycle

SUMMARY:
Evaluate the cardiovascular properties of MANP in AA with Hypertension

DETAILED DESCRIPTION:
The study is designed in 2 cycles.

Cycle 1 will incorporate 20 participants and include a screening / enrollment visit and 1 study visit. The study visit will be 30 hours and involves SQ administration of placebo (n=10) or MANP 2.5 ug/kg (n=10). Cycle 2 will incorporate 10 participants and include a screening / enrollment visit and 1 study visit. The study visit will be 30 hours and involves SQ administration of MANP 5 ug/kg (n=10). Studies will be performed at either the CRU of Mayo Clinic's CCaTS in Rochester, Minnesota or the University of Mississippi CRU in Jackson, Mississippi.

All participants will have a screening / enrollment visit where a medical history will be obtained and physical examination performed. At this visit informed consent will also be obtained. Hypertension validation as described above will follow. Once hypertension is validated, subjects will be scheduled for the study visit where either placebo or MANP will be administered at Mayo Clinic's or the University of Mississippi's CRU. Three days prior to the study visit, subjects will be initiated on a moderate sodium (3.0g/day) diet. Fluid intake will be restricted to 2.5 liters per day for all subjects. A 24-hour urine sodium collection will be obtained on the 24 hours prior to the study visit to establish adherence to the low sodium diet. Subjects will be maintained on their standard anti-HTN treatment for the entire duration of the study. At the study visit, subjects will be admitted at 07:00 to the CRU fasting. For safety purposes, all subjects will remain in the CRU a total of 24 hours following dosing. The study will be single blind.

Cycle 1:

At the study visit, either SQ placebo (n=10) or SQ MANP 2.5 ug/kg (n=10) will be administered.

Subjects will also be admitted at 07:00 to the CRU in the fasting state. Subjects will take their usual antihypertensive medications in the CRU at time "0 minutes". Over the next 60 minutes, blood pressure, heart rate, renal clearance, neurohumoral and cGMP assessment will be performed as outlined in Table 2. Ninety minutes after administration of the participant's usual antihypertensive medications, SQ placebo or SQ MANP will be administered if the systolic blood pressure is ≥ 120 mm Hg. Blood pressure and heart rate will be measured before and at several intervals after SQ placebo or SQ MANP administration. Four clearances of 6 hrs for total of 24 hrs after the dosing will be performed. At the end of each clearance, the patients will be asked to drink an amount of water equivalent to the sum of blood losses and urinary volume. During each clearance, urinary, hormonal, and hemodynamic measurements will be obtained and averaged for analysis. Subjects will be discharged from the CRU 24 hours after SQ placebo or SQ MANP administration.

If ≤2 study participants who received SQ MANP 2.5 μg/kg experience any of the adverse events listed below then cycle 2 will be initiated. If >2 study participants who received SQ MANP 2.5 μg/kg MANP experience one of the above events then the study will be terminated and we will not proceed to cycle 2.

* Clinically significant hypotension, defined as a decrease from baseline in clinical SBP ≥ 30 mmHg, or a decrease in sitting SBP to < 90 mmHg, or lightheadedness or dizziness or visual symptoms for 5 minutes.
* Any other safety results or adverse experiences that, in the opinion of the investigator, raise concerns about the safety or tolerability of a higher dose.

Cycle 2:

Cycle 2 will commence only if subjects in cycle 1 tolerated SQ MANP 2.5 μg/kg without clinically significant hypotension or other adverse events (as defined above).

In cycle 2, SQ MANP 5 ug/kg (n=10) will be administered at the study visit.

Subjects will also be admitted at 07:00 to the CRU in the fasting state. Subjects will take their usual antihypertensive medications in the CRU at time "0 minutes". Over the next 60 minutes, blood pressure, heart rate, renal clearance, neurohumoral and cGMP assessment will be performed as outlined in Table 2. Ninety minutes after administration of the participant's usual antihypertensive medications, SQ MANP will be administered if the systolic blood pressure is ≥ 120 mm Hg. Blood pressure and heart rate will be measured before and at several intervals after SQ placebo or SQ MANP administration. Four clearances of 6 hrs for total of 24 hrs after the dosing will be performed. At the end of each clearance, the patients will be asked to drink an amount of water equivalent to the sum of blood losses and urinary volume. During each clearance, urinary, hormonal, and hemodynamic measurements will be obtained and averaged for analysis. Subjects will be discharged from the CRU 24 hours after SQ placebo or SQ MANP administration.

ELIGIBILITY:
Inclusion Criteria:

1. Hypertension, defined as a mean supine BP equal to or greater than 140 mmHg and taking at least one standard of care therapies (including a diuretic, angiotensin converting enzyme inhibitor or angiotensin receptor blocker and a calcium channel blocker);
2. MDRD estimated GFR > 30 mL/min to be calculated at the screening visit by available serum creatinine
3. Male or female African Americans
4. Have a body mass index (BMI) within the range of 18-40 kg/m2;
5. Be able to communicate effectively with the study personnel
6. Be adequately informed of the nature and risks of the study and give written informed consent prior to receiving study medication.

Exclusion Criteria:

1. Known hypersensitivity or allergy to MANP or other NPs;
2. Women of child bearing age
3. Having received any investigational drug or device within 30 days prior to entry into the study; 4) A history (within the last 2 years) of alcohol abuse, illicit drug use, significant mental illness, physical dependence to any opioid, or any history of drug abuse or addiction;
4. A history of difficulty with donating blood or donated blood or blood products within 45 days prior to enrollment;
5. Clinically significant new illness in the 1 month before screening in the opinion of the investigator;
6. History of severe allergies;
7. History of CAD, CVD or syncope;
8. History of epilepsy or other seizure disorder;
9. History of organ transplantation;
10. Malignancy within 5 years;
11. Clinically significant intrinsic renal disease, renal artery stenosis, or history of fibromuscular dysplasia of the renal arteries and;
12. Consumption of a phosphodiesterase-5 inhibitor.
13. Known adrenal insufficiency
14. Subjects with orthostatic hypotension at the screening visit, defined as a decrease in systolic BP of >20 mmHg or a decrease in diastolic BP of >10 mmHg within three minutes of standing when compared with blood pressure from the sitting position.
15. Subjects with a systolic BP >180 mmHg or a diastolic BP >100 mmHg while sitting

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Blood Pressure | 12 hours
  The primary outcome is change in blood pressure 12 hours after MANP or placebo administration compared to the baseline blood pressure. Blood pressure will be measured by an automated arm blood pressure cuff. The unit of measurement is mm Hg. Time frame = 12 hours.

SECONDARY OUTCOMES:
Urinary cGMP excretion | 12 hours
  Urinary cGMP excretion (pmol/min) 12 hours after MANP or placebo administration compared to baseline measurement. Urinary cGMP excretion will be measured by a 30 minute urine collection.
Urinary sodium excretion | 12 hours
  Urinary sodium excretion (mEq/min) 12 hours after MANP or placebo administration compared to baseline measurement. Urinary sodium excretion will be measured by a 30 minute urine collection.
Glomerular filtration rate | 12 hours
  Glomerular filtration rate (ml/min) 12 hours after MANP or placebo administration compared to baseline measurement. GFR describes the flow rate of filtered fluid through the kidney measured in milliliters per minute per 1.73 m^2 of body surface area and will be determined by iothalamate clearance.
Plasma aldosterone | 12 hours
  Plasma aldosterone 12 hours after MANP or placebo administration compared to baseline measurement. Aldosterone is measured by analyzing a blood specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Paul M McKie, M.D., Principal Investigator — Mayo Foundation
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials